CLINICAL TRIAL: NCT03269890
Title: The Efficacy of Intermediate Cervical Plexus Block Versus Cutaneous and Thyroid Capsular Blocks in Thyroid Surgeries
Brief Title: The Efficacy of Intermediate Cervical Plexus Block Versus Cutaneous and Thyroid Capsular Blocks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: MS/17.03.138
Record Dates: First submitted 2017-08-29; First posted 2017-09-01 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Thyroid Surgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Capsule and cutaneous blocks (Experimental): 7.5 mL of 0.5% bupivacaine + Epinephrine 5 ug/ ml for both blocks per side. once before surgery
  Interventions: Procedure: Capsule and cutaneous blocks
- US-intermediate cervical plexus block (Active Comparator): 15 mL of 0.5% isobaric bupivacaine + Epinephrine 5 microgram/ ml. per side. once before surgery
  Interventions: Procedure: US-intermediate cervical plexus block

INTERVENTIONS:
Procedure: Capsule and cutaneous blocks — 7.5 mL of 0.5% bupivacaine + Epinephrine 5 ug/ ml for both blocks once before surgery per side
  Arms: Capsule and cutaneous blocks
Procedure: US-intermediate cervical plexus block — 15 mL of 0.5% bupivacaine + Epinephrine 5 ug/ ml once before surgery per side.
  Arms: US-intermediate cervical plexus block

SUMMARY:
Thyroid gland surgery is one of the most commonly performed operations for either benign or malignant pathologies Pain related to thyroid surgery is of moderate intensity .which may be treated with NSAIDs or opioids. However, Opioids have many well-known undesirable effects, including postoperative nausea and vomiting, which are frequent after this type of procedure.

DETAILED DESCRIPTION:
Regional techniques of anesthesia may help to decrease post-operative pain and reduce systemic analgesic requirement. Classically, the cervical plexus is considered to have two distributions, the superficial cutaneous and the deep motor nerves.

Anatomically, the thyroid gland has an inner true capsule which is thin and adheres closely to the thyroidal tissue [Fancy et al., 2010]. External to this is a false capsule formed by the middle layer of the deep cervical fascia, which splits anterolaterally to ensheathe the thyroid gland, thus forming the thyroid sheath [Bliss et al., 2000]. In this fashion, the potential space called the capsule-sheath space is formed. It contains also loose connective tissue, blood vessels, nerves and parathyroid gland. Anesthetic deposited in this space would block the surface of thyroid gland and permeate directly into the parenchyma producing effective local anesthesia for thyroid surgical procedures. It is supposed also to involve autonomic nerve block of the thyroid gland [Fliers et al., 2010]. Additionally, a subcutaneous injection along the sternocleidomastoid muscle (SCM) would also enhance effective local anesthesia for the initial skin incision and further contribute to a more ideal working environment for the surgeon. Therefore, anesthetic technique termed ultrasound-guided capsule-sheath space block (CSSB) combined with anterior cervical cutaneous nerves block (CCNB) for thyroidectomy is done [Wang et al., 2015] .

Our hypothesis is that a combination of simple dual techniques including superficial cutaneous block to provide sensory blockade, and surgeon mediated capsular block may afford autonomic thyroid blockade. In comparison, ultrasound guided intermediate cervical plexus block may provide these blocks but using a machine and deep penetration possibly involving unwanted blocks for phrenic and recurrent laryngeal nerves. So, if the simple safe technique can provide the same intra and postoperative anesthetic conditions it will be preferred.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status grade I and grade II.
* Euthyroidism after thyroid function tests

Exclusion Criteria:

* Patient refusal.
* Thyroid gland more than 5 cm size.
* Retrosternal extension.
* Planned block neck dissection.
* Neuromuscular diseases
* Hematological diseases.
* Bleeding diseases.
* Coagulation abnormality.
* Psychiatric diseases.
* Drug abuse.
* Local skin infection
* sepsis at site of the block.
* Known intolerance to the study drugs.
* Body Mass Index > 40 Kg/m2.
* Known diaphragmatic motion abnormalities
* major respiratory disease.
* Previous history of cervical surgery.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Total dose of opioid analgesics used | For 24 hours after surgery
  The total dose of opioid analgesics required in the post-operative periods

SECONDARY OUTCOMES:
Postoperative pain | For 24 hours after surgery
  Postoperative visual analogue score (VAS) (0 no pain -10 worst imaginable pain),
Time to first analgesic request | For 24 hours after surgery
  Time to first request for a rescue analgesic
Fentanyl use | For 5 hours after start of anaesthesia
  Intraoperative use of fentanyl
Rocuronium use | For 5 hours after start of anaesthesia
  Intraoperative use of rocuronium
Sensory blockade | for 1 hour after surgery
  Assessment of sensory blockade
Diaphragmatic dysfunction | for 5 hours after performing blockade
  Diaphragmatic dysfunction using ultrasound assessment and possible x ray
Sedation score | for 5 hours after performing blockade
  Sedation score using Modified Ramsay scale
Patient satisfaction | for 24 hrs after surgery
  Patient satisfaction regards analgesia using a score of (0-10) with 10 represents the highest satisfaction
Postoperative nausea and vomiting | For 24 hours after surgery
  frequency
Postoperative headache | For 24 hours after surgery
  frequency
Hoarseness of voice | For 24 hours after surgery
  frequency
Dysphagia | For 24 hours after surgery
  frequency
Respiratory difficulty | For 24 hours after surgery
  Peripheral oxygen saturation less than 92%

CONTACTS AND LOCATIONS:
Overall Officials: Moneir O El-Hefny, MD, Study Chair — Professor of Anesthesia and Surgical Intensive Care
Locations (1):
- Oncolgy Center, Mansoura University,, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: Undecided